CLINICAL TRIAL: NCT05828173
Title: PINNACLE I Clinical Study: a Clinical Trial to Assess the Elixir Medical LithiX Coronary Hertzian Contact Intravascular Lithotripsy Catheter for Treatment of Moderately to Severely Calcified, Stenotic De Novo Coronary Artery Lesions
Brief Title: A Clinical Trial to Assess the Elixir Medical LithiX Coronary Hertzian Contact Intravascular Lithotripsy Catheter
Acronym: PINNACLE-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-2202
Record Dates: First submitted 2023-04-03; First posted 2023-04-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Lithotripsy, Calcified Coronary Lesions
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LithiX Coronary Hertzian Contact Intravascular Lithotripsy Treatment (Experimental)
  Interventions: Device: LithiX Coronary Hertzian Contact Intravascular Lithotripsy Catheter (LithiX Coronary HCIVLC; LithiX)

INTERVENTIONS:
Device: LithiX Coronary Hertzian Contact Intravascular Lithotripsy Catheter (LithiX Coronary HCIVLC; LithiX) — Vessel preparation of moderately to severely calcified coronary artery lesions prior to stenting allows for full stent expansion and apposition to the vessel wall

SUMMARY:
The objective of the PINNACLE I Clinical Study is to assess safety and performance of the LithiX Coronary Hertzian Contact Intravascular Lithotripsy Catheter (LithiX Coronary HCIVLC; LithiX) to treat moderately to severely calcified coronary artery lesions by calcium fragmentation utilizing Hertzian contact stress from LithiX HCIVLC.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single-arm clinical study. Enrollment of up to 60 patients requiring percutaneous coronary intervention (PCI) on up to two de novo coronary artery lesions with reference vessel diameters ≥ 2.25 mm and ≤ 3.5 mm, and lesion lengths of ≤ 34 mm, with moderate to severe calcification.

The LithiX Coronary HCIVLC is a proprietary Hertzian contact intravascular lithotripsy catheter delivered through the coronary arterial system to visualize and treat calcified stenoses potentially resistant to full stent expansion. The LithiX Coronary HCIVLC consists of a semi-compliant balloon featuring multiple rows of stainless-steel hemispheres which are intended to atraumatically fragment calcium via Hertzian contact intravascular lithotripsy.

In the Optical Coherence Tomography (OCT) imaging subgroup, approximately 30 patients will undergo OCT imaging at pre-procedure, post-LithiX treatment, and the end of procedure following stent deployment.

Subjects will be followed through hospital discharge and will have clinical follow-up conducted by phone at 30 days and 6 months post-index procedure.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedures.
3. Subject must agree not to participate in any other clinical study during the course of the study that would interfere with the endpoints of this study.
4. Subjects must have a single or double vessel coronary artery disease (CAD) and clinical evidence of ischemic heart disease, such as CAD, silent ischemia, stable / unstable angina, and NSTEMI if biomarkers are stable or falling at time of inclusion.

Angiographic Inclusion Criteria:

1. Subject must have de novo lesion(s) in native coronary arteries suitable for percutaneous coronary intervention.
2. Up to 2 de novo coronary artery lesions in separate epicardial vessels, which are moderately to severely calcified, meeting all of the following criteria visually assessed by angiography:

   * ≥70% diameter stenosis by visual estimation
   * reference vessel diameters of 2.25 mm - 3.5 mm
   * lesion length of ≤ 34 mm
   * TIMI flow ≥ 1 at baseline
3. Any non-target lesion must be located in different coronary artery from a target lesion. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion and must be deemed a clinical angiographic success as visually assessed by the physician.

General Exclusion Criteria:

1. Subject with a known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, anti-platelet medications, or sensitivity to contrast media which cannot be adequately pre-medicated.
2. Subject with known diagnosis of STEMI at index presentation or within 7 days of study screening.
3. Patient refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery.
4. Subject with known pregnancy or is nursing. Women of child-bearing potential should have a documented negative pregnancy test within 7 days before index procedure.
5. Planned use of atherectomy, laser, lithoplasty, thrombectomy, scoring or cutting balloon, or any investigational device other than LithiX in the target lesion during the index procedure.
6. Patients on renal dialysis or with known eGFR < 30 ml/min.
7. NYHA class III or IV heart failure.
8. Patient has active systemic infection.
9. Cerebrovascular accident (CVA) or transient ischemic attach (TIA) within the past 6 months.
10. Active peptic ulcer or active gastrointestinal (GI) bleeding within the past 6 months.
11. Subject has a known left ventricular ejection fraction (LVEF) <30% (LVEF may be obtained at the time of the index procedure if the value is unknown, if necessary).
12. Subject is a member of a vulnerable population as defined GCP E6, including individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Angiographic Exclusion Criteria:

1. More than two target lesions or more than 1 target and 1 non-target lesion requiring treatment.
2. Extreme angulation (90º or greater) proximal to or within the target lesion.
3. Previous percutaneous intervention of lesions in a target vessel (including side branches) conducted within 6 months before the study procedure, or any prior lesion treated within 10 mm (proximal or distal) from the current target lesion.
4. Previous percutaneous intervention of lesions in a non-target vessel (including side branches) conducted within 30 days before the study procedure.
5. Angiographic evidence of a target lesion dissection prior to LithiX Hertzian Contact Lithotripsy.
6. Visible thrombus (by angiography) at target lesion site.
7. Unprotected left main coronary artery disease (Greater than 50% diameter stenosis).
8. Target lesion is located in a native vessel distal to anastomosis with a saphenous vein graft or LIMA/RIMA bypass.
9. Evidence of aneurysm in target vessel.
10. Coronary artery spasm of the target vessel in the absence of a significant stenosis.
11. Target lesion involves a bifurcation requiring treatment with more than one stent or pre-dilatation of a side branch >2.0 mm in diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Clinical success | At the end of procedure
  This is the primary effectiveness and safety endpoint and defined as residual stenosis <50% after final treatment (with or without stenting) with no evidence of in-hospital major adverse cardiovascular events (MACE).
Major adverse cardiovascular events (MACE) | 30 days
  This is the primary safety endpoint and defined as a per-subject composite endpoint of cardiovascular death, myocardial infarction, and target vessel revascularization.

SECONDARY OUTCOMES:
Angiographic success | During the procedure
  defined as success in facilitating stent delivery with <50% residual stenosis and without serious angiographic complications
Optical Coherence Tomography (OCT) imaging | During the procedure
  assessment of the lesion and stent in a subset of patients
All myocardial infarction | Through study completion, an average of 6 months
  Q-wave and non-Q-wave
Target vessel revascularization | Through study completion, an average of 6 months
  defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel including the target lesion.
Target lesion revascularization | Through study completion, an average of 6 months
  defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion
Target lesion failure | Through study completion, an average of 6 months
  defined as a per-subject composite endpoint of cardiovascular death, target vessel myocardial infarction, and clinically-indicated target lesion revascularization
Stent thrombosis | Through study completion, an average of 6 months
  definite and probable stent thrombosis
All-cause death | Through study completion, an average of 6 months
  Cardiovascular and non-cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, PhD, Principal Investigator — ZNA Middelheim, Antwerp, Belgium; Johan Bennett, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen Leuven, Leuven, Belgium
Locations (7):
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Ziekenhuis Oost-Limburg, Campus Sint Jan, Genk
  - Jessa Ziekenhuis, Hasselt
  - Universitaire Ziekenhuizen Leuven, Leuven
- Netherlands (3):
  - Meander Medical Centre, Amersfoort
  - Catharina Ziekenhuis, Eindhoven
  - Maasstad Ziekenhuis, Rotterdam

IPD SHARING:
Plan to Share IPD: No